CLINICAL TRIAL: NCT00731289
Title: Efficacy and Safety of Intra-Articular Injections of Durolane® in the Treatment of Osteoarthritis in the Knee
Brief Title: Gait Patterns After Intraarticular Treatment of Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: University Hospital Muenster (Other)
Responsible Party: Adrian Skwara, Department of Orthopaedics and Rheumatology, University Hospital Marburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3II Fuchs
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Knee; Hyaluronan; Gait Analysis
MeSH Terms: conditions — Osteoarthritis | interventions — Hyaluronic Acid; Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): single intraarticular injection of hyaluronan 3 ml (Durolane®, 20 mg/ml non-animal stabilized hyaluronic acid (NASHA) in buffered physiological sodium chloride solution pH 7 in one pre-filled glass syringe in sterile pack
  Interventions: Drug: hyaluronic acid
- 2 (Active Comparator): single intraarticular injection of triamcinolone 1 ml (Volon A10®, 10mg triamcinolone acetonide, 10mg/ml)
  Interventions: Drug: triamcinolone

INTERVENTIONS:
Drug: hyaluronic acid — one intraarticular injection of hyaluronan (HA) 3 ml (Durolane®, 20 mg/ml non-animal stabilized hyaluronic acid (NASHA) in buffered physiological sodium chloride solution pH 7 in one pre-filled glass syringe in sterile pack
  Other Names: 20 mg/ml non-animal stabilized hyaluronic acid (NASHA)
  Arms: 1
Drug: triamcinolone — one intraarticular injection of triamcinolone 1 ml (Volon A10®, 10mg triamcinolone acetonide, 10mg/ml)
  antiinflammatory intervention
  Other Names: triamcinolone acetonide, 10mg/ml
  Arms: 2

SUMMARY:
The aim of this study was to analyse the difference of the functional and clinical outcome after intraarticular treatment of patients with osteoarthritis of the knee with a single injection of hyaluronan (HA) or Triamcinolone (TA) with respect to the quality of life during the study period.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common chronic joint disease of the aging patient. The primarily affected joints are the knee and hip. The progress of the disease has an important influence on the patient´s life, including functional and social activities, body image and emotional well being. Furthermore, socioeconomic aspects play an eminent role in the treatment of osteoarthritis in joints.

In non-operative treatment, pain reduction and improved function are the primary goals. It is important to distinguish between systemic and local therapeutic options. In the systemic treatment, palliation of pain can be achieved by simple analgetics, non- steroidal anti-inflammatory drugs and opioids. Local therapy can selectively treat the symptomatic joint. Intraarticular application of different drugs by injection can be performed. Glucocorticoids are the most commonly used intraarticular agents, which reduce pain and improve function and well being. In recent years, the intraarticular use of different hyaluronan (HA) products became more widely accepted. Hyaluronan is a physiological component of the synovial fluid and cartilage matrix. It is responsible for the viscoelastic properties of the synovial fluid. In osteoarthrotic joints, the molecular weight and the concentration of endogenous HA are decreased compared with healthy joints. This implies a reduction of the viscoelasticity of the synovial fluid. In order to restore this viscoelasticity, augment the flow of the synovial fluid, normalise the synthesis and inhibit the degradation of endogenous hyaluronan, an application of exogenous HA can be performed. The therapeutic effects and the safety of intraarticular application of HA in the treatment of OA in the knee have been demonstrated in several clinical trials. Until now there are only three studies that objectively analysed few aspects of the functional outcome after treatment with HA.

ELIGIBILITY:
Inclusion Criteria:

* men and women between 35 and 80 years of age
* radiographically verified degenerative osteoarthritis of the knee (grade II or III according to the Kellgren and Lawrence classification)
* pain of at least 40 mm on a 100 mm visual analogue scale (VAS) at initial examination
* persisting pain for at least 6 months
* Lequesne-Score of at least 10 points
* good physical and mental status
* good compliance and agreement to participate in this study

Exclusion Criteria:

* non-degeneratively induced osteoarthritis
* rheumatoid arthritis
* ligamentous instability or complete resection of the meniscus
* Sudeck´s disease
* operations of the affected knee within the last three months
* varus or valgus deformity of more than 15 degrees
* patellofemoral arthritis
* intraarticular therapy of the affected joint within the last 6 months with hyaluronan and three months with glucocorticoids
* severe systemic diseases (tumor, exacerbated diabetes mellitus, hyperthyroidism)
* anti-thrombotic medication or regular medication with NSAID/psychiatric pharmaceuticals
* infectious diseases
* alcohol abuse
* drugs
* psychiatric diseases or suicidal tendencies
* involvement in another study
* non-compliance
* acute hemarthrosis or joint effusion
* allergic predisposition
* skin infections or skin diseases around the knee

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
visual analogue scale for pain (VAS) | 12 weeks

SECONDARY OUTCOMES:
gait analysis | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Fuchs-Winkelmann, Prof. MD, Study Chair — University Hospital Marburg
Locations (1):
- Department of Orthopaedics, Movement Analysis Lab, University Hospital Münster, Germany, Münster, Germany